CLINICAL TRIAL: NCT06563960
Title: Effect of Carbonated Water on Swallowing in Patients With Liquid Dysphagia
Brief Title: Effect of Carbonated Water on Swallowing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, Clinical Professor, Federal University of Health Science of Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: carbonated water
Record Dates: First submitted 2024-06-01; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Carbonated Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Other): patients who drank carbonated water.
  Interventions: Other: carbonated water

INTERVENTIONS:
Other: carbonated water — Participants will drink carbonated water during videofluoroscopy.

SUMMARY:
Swallowing has an important function in the lives of individuals, it is related to moments of socialization, pleasure, nutrition and also helps protect against the entry of food, saliva or other material towards the lungs (penetration and/or laryngotracheal aspiration). A Difficulty in swallowing is called dysphagia and therapeutic strategies are necessary to help the affected individuals. The use of carbonated water as a therapeutic strategy has been used, however, there are still few studies on the topic. In the search for therapeutic strategies viable and easy to insert into the clinical routine and daily lives of patients, this study aims to verify the effect of carbonated water on swallowing liquids for patients with dysphagia diagnosed by videodeglutogram examination, through comparison with non-water carbonated. The present study aims to generate scientific evidence about the effect of water carbonated drink as a strategy in patients with liquid dysphagia, with the aim of helping professional speech therapist and other professionals involved in the therapeutic process, in order to improve the health and quality of life of dysphagic patients and contribute to the evolution of knowledge in the field of dysphagia. This is a clinical trial, all participants will be included adult patients to carry out the video swallow examination, which present aspiration and/or laryngotracheal penetration of liquids during the performance of the and who agree to participate in the research. The effect of carbonated water on levels of penetration and/or laryngotracheal aspiration in relation to the use of non-carbonated water, and analyzed whether the results obtained with the use of carbonated water have behavior similar between the different patient profiles studied.

DETAILED DESCRIPTION:
This is a clinical trial. The study population comprises all adult dysphagic patients who present laryngotracheal penetration and/or aspiration of liquids during the videodeglutogram exam, performed at the aforementioned Imaging Diagnosis Center, during the period from March to December 2023 and who agree to participate. Therefore, a convenience sample will be used.

The study population will consist of all patients who present laryngotracheal penetration and/or aspiration of liquids during the videodeglutogram exam performed at the institution's Imaging Diagnosis Center and who agree to participate in the study. The anamnesis was constructed by the research team, aiming to collect information about the target population (age, sex, marital status, education, underlying pathology, main complaint and swallowing difficulties). In addition, for those who have a history in the electronic medical record, the same will be consulted to verify information regarding the history of previous illnesses, medications in use and general health conditions. The examination will be performed by the technically responsible speech therapist, with experience in the area. It consists of offering food to the patient (thin liquid - water, moderately thickened - yogurt, soft solid - bread and hard - crackers), impregnated with a barium contrast; during swallowing, dynamic, real-time images are captured by an x-ray equipment, making it possible to evaluate all phases of swallowing, following the path of the food from the mouth to the stomach. The following aspects will be checked: oral preparation of the food, ejection of the bolus, the existence of early food escape and identification of the location of the beginning of the pharyngeal phase of swallowing, the presence of stasis in valleculae and pyriform sinuses, episodes of laryngotracheal penetration and/or aspiration, and changes in esophageal motility. Some compensatory strategies, such as head positioning and airway protection maneuvers, may be tested during the examination. Patients who present laryngotracheal penetration and/or aspiration with thin liquid will be subjected to the ingestion of carbonated water in order to verify whether there will be a change in the pattern of laryngotracheal penetration and/or aspiration. The carbonated water chosen for the study was the brand; for every 60ml of water, 1.8ml of barium (3% concentration) will be mixed, the contrast required for the images to be captured in the videofluoroscopy examination. To classify the functional severity of dysphagia and describe laryngotracheal penetration and/or aspiration, the following scales will be considered: Dysphagia Outcome and Severity Scale (DOSS) and Rosenbek Scale. The classification for evaluating the biomechanics of swallowing will be made based on the results of the videofluoroscopy exam, which will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 18 years old;
2. Individuals who present penetration and/or laryngotracheal aspiration for liquids during the video swallow examination.

Exclusion Criteria:

1. Patients with contraindication to liquid testing (those with evidence of massive aspiration of moderately thickened food where it is necessary to interrupt examination per safety protocol, who have previously had a tracheoesophageal fistula diagnosed or who do not present any swallowing response);
2. Individuals who present clinical instability and sensory oscillation that make it impossible to carrying out the exam;
3. Individuals who present postural changes that limit positioning for carrying out the exam;
4. Patients who are allergic to barium contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who reduce or eliminate penetration and/or aspiration with carbonated water. | 12 months
  Check for how many participants this strategy is effective in reducing penetration and/or aspiration.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fabricio Edler Macagnan, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No